CLINICAL TRIAL: NCT06672120
Title: Exercise in Regional Breast Cancer With Neoadjuvant Anthracycline- Based Chemotherapy and Immunotherapy With Checkpoint-Inhibition
Brief Title: Exercise in Triple- Negative Breast Cancer
Acronym: ExACT-ICI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024-396-S-KK
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Cancer, Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with TNBC and scheduled for immuno-chemotherapy will be randomized (1:1) into an intervention group receiving combined endurance and resistance training and a control group receiving standard exercise recommendations.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal investigator, who will assess outcomes, will be blinded to group allocation. Patients will be randomized by a staff member. Data analysis will be done by a professional statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive home-based, video-supervised exercise training from a sports scientist. Training will consist of elements of moderate continuous and high-intensity endurance training as well as resistance training.
  Interventions: Behavioral: Exercise training
- Control Group (No Intervention): The control group will receive standard recommendations on physical activity.

INTERVENTIONS:
Behavioral: Exercise training — Combined, home-based, supervised, video- assisted, endurance and resistance training
  Arms: Intervention Group

SUMMARY:
This is a prospective, randomized, controlled mono-center study investigating the effects of a combined, supervised aerobic exercise and resistance training in female patients with newly diagnosed, therapy-naive triple-negative breast cancer (TNBC, stage I-III) between 18 and 50 years of age scheduled for anthracycline-based chemotherapy and immunotherapy with checkpoint inhibitors. All patients will receive smart watches for rhythm monitoring.

Patients will be randomized (1:1) into a control group, receiving 24 weeks of standard exercise recommendations during neoadjuvant therapy, and an intervention group receiving 24 weeks of home-based, video-supervised exercise training consisting of endurance and resistance training. The primary endpoint is the change of peak oxygen consumption (VO2peak) between baseline and 24 weeks in the groups. Secondary endpoints include changes of physical function (short physical performance battery, SPPB), as well as cardiac biomarkers, quality of life, and changes of strength of the upper and lower body between baseline and 24 weeks. In addition, variables of cardiopulmonary exercise testing (CPET), resting and stress echocardiography, and burden of atrial fibrillation (AF) will be assessed. All changes in variables will be analyzed from baseline until 52 weeks as well.

Both groups will receive standard exercise recommendations after 24 weeks and will be followed-up by clinical examination after 52 weeks. Echocardiographic variables (at rest and during exercise), quality of life, CPET, SPPB, strength testing, burden of AF, and cardiac biomarkers will be assessed. Changes between the end of the intervention period 24 weeks after diagnosis and the end of follow-up after 52 weeks will be analyzed. In addition, changes in variables between baseline and 52 weeks will be analyzed.

As an exploratory endpoint the incidence of cancer therapy-related cardiac dysfunction (CTRCD) and immune-checkpoint inhibitor- associated myocarditis (ICI-myocarditis) will be assessed after 24 and 52 weeks.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled mono-center study investigating the effects of a combined, supervised aerobic exercise and resistance training in female patients with newly diagnosed TNBC (stage I-III) between 18 and 65 years of age scheduled for anthracycline-based chemotherapy and immunotherapy with checkpoint inhibitors. All patients will receive smart watches for rhythm monitoring. Patients will be advised to trigger electrocardiogram (ECG) measurements every day at 8 a.m., 2 p.m. and 8 p.m. as well as before and immediately after every training session (intervention group only). In addition, ECG should be recorded whenever symptoms occur.

Patients will be randomized (1:1) into a control group, receiving 24 weeks of standard exercise recommendations during neoadjuvant therapy, and an intervention group receiving 24 weeks of home-based, video-supervised exercise training consisting of endurance and resistance training.

At baseline clinical examination, quality of life, cardiac biomarkers, resting and stress echocardiography and CPET will be performed. SPPB and strength of the upper and lower body will be assessed.

Training in the intervention group will be performed 5x/week with 20 minutes/session and will contain resistance training and endurance training as a mixture between moderate continuous and high-intensity interval training. Training corridors based on heart rate will be prescribed with the aid of CPET testing at baseline and during follow-up visits. Intensity will be progressively increased, but will be individually adapted to the schedule and response to chemo- and immunotherapy.

Follow-up visits will be performed six and twelve weeks after diagnosis and clinical examination, cardiac biomarkers, resting and stress echocardiography and CPET as well as testing of muscle strength, SPPB, and quality of life will be repeated. Prescribed training corridors of heart rate will be adapted after each test. Upon clinical suspicion for adverse events, such as ICI-myocarditis, magnetic resonance imaging of the heart will be performed and training will not be continued.

The primary endpoint is the change of VO2peak between baseline and 24 weeks in the groups. Secondary endpoints include changes of variables between baseline and 24 weeks, including SPPB, cardiac biomarkers, quality of life, changes of strength of the upper and lower body (knee extensor and biceps muscles), variables of CPET, resting and stress echocardiography, and burden of AF. Changes in variables between baseline and after 52 weeks will also be analyzed. 24h- Holter monitoring will be performed at the end of weeks 24 and 52.

Both groups will receive standard exercise recommendations after 24 weeks and will be followed-up by clinical examination after 52 weeks: Resting and stress echocardiography, quality of life, CPET, SPPB, strength testing, AF burden, and cardiac biomarkers will be re-assessed.

As an exploratory endpoint the incidence CTRCD and ICI-myocarditis will be assessed after 24 and 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with newly diagnosed, local triple-negative breast cancer (stage I-III) ≥ 18 to 65 years of age scheduled for immunochemotherapy with pembrolizumab and anthracycline-based chemotherapy

Exclusion Criteria:

* Unstable cardiac condition (clinical suspicion of progress or unstable coronary artery disease, signs of acute heart failure, haemodynamically relevant arrhythmias)
* Orthopaedic disability to exercise

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer patients as defined by the treating gynaecologist
Enrollment: 120 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen consumption (VO2peak) from baseline until the end of intervention | 24 weeks
  Difference of VO2peak between baseline to the end of intervention per group

SECONDARY OUTCOMES:
VO2peak from baseline to the end of follow-up | 52 weeks
  Difference of VO2peak between baseline to the end of follow-up per group
VO2peak from the end of intervention to the end of follow-up | 28 weeks
  Difference of VO2peak between the end of intervention and the end of follow-up per group
Burden of atrial fibrillation (AF) from baseline to the end of intervention | 24 weeks
  Burden of AF will be assessed with 24h-Holter monitoring at the end of week 24 and with patient-triggered documentation through smart watch monitoring. ECG triggering will be done every day throughout the study at 8 a.m., 2 p.m., 8 p.m., before and immediately after exercise, or with perceived symptoms
Burden of AF from baseline to the end of follow-up | 52 weeks
  Burden of AF will be assessed with 24h-Holter monitoring at the end of week 24 and 52 and with patient-triggered documentation through smart watch monitoring. ECG triggering will be done every day throughout the study at 8 a.m., 2 p.m., 8 p.m., before and immediately after exercise, or with perceived symptoms
Burden of AF from the end of intervention to the end of follow-up | 28 weeks
  Burden of AF will be assessed with 24h-Holter monitoring at the end of week 24 and 52 and with patient-triggered documentation through smart watch monitoring. ECG triggering will be done every day throughout the study at 8 a.m., 2 p.m., 8 p.m., before and immediately after exercise, or with perceived symptoms
Performance in short physical performance battery (SPPB) from baseline to end of intervention | 24 weeks
  Values range from 0 (worst performance) to 12 (best performance)
Performance in SPPB from the end of intervention to the end of follow-up | 28 weeks
  Values range from 0 (worst performance) to 12 (best performance)
Performance in SPPB from baseline to the end of follow-up | 52 weeks
  Values range from 0 (worst performance) to 12 (best performance)
Improvement of muscle strength of the upper (biceps curl) and lower extremity (knee extensor) from baseline to the end of intervention | 24 weeks
  A one repetition maximum test (1 RPM) will be done for both tests
Improvement of muscle strength of the upper (biceps curl) and lower extremity (knee extensor) from baseline to the end of follow-up | 52 weeks
  1 RPM will be done for both tests
Improvement of muscle strength of the upper (biceps curl) and lower extremity (knee extensor) from the end of intervention to the end of follow-up | 28 weeks
  1 RPM will be done for both tests
Changes of resting and stress echocardiographic variables from baseline to the end of intervention | 24 weeks
  Left ventricular ejection fraction will be measured at rest and peak exercise
Changes of resting and stress echocardiographic variables from baseline to the end of follow-up | 52 weeks
  Left ventricular ejection fraction will be measured at rest and peak exercise
Changes of resting and stress echocardiographic variables from the end of intervention to the end of follow-up | 28 weeks
  Left ventricular ejection fraction will be measured at rest and peak exercise
Cardiac biomarkers from baseline to the end of intervention | 24 weeks
  Change in troponin I and NTproBNP from baseline to the end of intervention
Cardiac biomarkers from the end of intervention to the end of follow-up | 28 weeks
  Change in troponin I and NTproBNP from the end of intervention to the end of follow-up
Cardiac biomarkers from baseline to the end of follow-up | 52 weeks
  Change in troponin I and NTproBNP from baseline to the end of follow-up
Change in quality of life from baseline to the end of intervention | 24 weeks
  Change in EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire). Values range from 0 to 100, with 100 showing the best quality of life and 0 the worst.
Change in quality of life from the end of intervention to the end of follow-up | 28 weeks
  Change in EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire). Values range from 0 to 100, with 100 showing the best quality of life and 0 the worst.
Change in quality of life from baseline to the end of follow-up | 52 weeks
  Change in EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire). Values range from 0 to 100, with 100 showing the best quality of life and 0 the worst.
Incidence of immune-checkpoint inhibitor associated myocarditis (ICI-myocarditis) from baseline to the end of follow-up | 52 weeks
  ICI myocarditis is defined as signs of myocarditis on magnetic resonance imaging of the heart according to the modified Lake Louis criteria and positive troponin I levels or positive troponin levels and two additional side criteria (clinical symptoms, reduction in left ventricular ejection fraction, strain, or wall motion abnormalities, or other immune-related side effects, or arrhythmias)
Decrease of minute ventilation to carbon dioxide production (VE/VCO2) from baseline to the end of intervention | 24 weeks
  Change in VE/VCO2 during CPET
Decrease of VE/VCO2 from baseline to the end of follow-up | 52 weeks
  Change in VE/VCO2 during CPET
Decrease of VE/VCO2 from the end of intervention to the end of follow-up | 28 weeks
  Change in VE/VCO2 during CPET
Incidence of cancer treatment-related cardiac dysfunction (CTRCD) from baseline to the end of follow-up | 52 weeks
  CTRCD is defined as a reduction of left ventricular ejection fraction ≥10% to 40-49% OR a reduction of <10% to 40-49% AND a decline of strain >15% of the baseline OR a new rise cardiac biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Simon Wernhart, MD, Principal Investigator — Technical University of Munich
Locations (2):
- Germany (2):
  - Preventive Sports Medicine and Sports Cardiology, Munich, Bavaria
  - Department of Medicine, Division of Prevention and Sports Medicine TU Munich, Munich

IPD SHARING:
Plan to Share IPD: No
Information can be attained from the principal investigator Simon Wernhart on reasonable request

REFERENCES:
- [Background] Lyon AR, Lopez-Fernandez T, Couch LS, Asteggiano R, Aznar MC, Bergler-Klein J, Boriani G, Cardinale D, Cordoba R, Cosyns B, Cutter DJ, de Azambuja E, de Boer RA, Dent SF, Farmakis D, Gevaert SA, Gorog DA, Herrmann J, Lenihan D, Moslehi J, Moura B, Salinger SS, Stephens R, Suter TM, Szmit S, Tamargo J, Thavendiranathan P, Tocchetti CG, van der Meer P, van der Pal HJH; ESC Scientific Document Group. 2022 ESC Guidelines on cardio-oncology developed in collaboration with the European Hematology Association (EHA), the European Society for Therapeutic Radiology and Oncology (ESTRO) and the International Cardio-Oncology Society (IC-OS). Eur Heart J. 2022 Nov 1;43(41):4229-4361. doi: 10.1093/eurheartj/ehac244. No abstract available. PMID 36017568
- [Result] Wernhart S, Rassaf T. Relevance of Cardiovascular Exercise in Cancer and Cancer Therapy-Related Cardiac Dysfunction. Curr Heart Fail Rep. 2024 Jun;21(3):238-251. doi: 10.1007/s11897-024-00662-0. Epub 2024 May 2. PMID 38696059
- [Result] Wernhart S, Rassaf T. Exercise, cancer, and the cardiovascular system: clinical effects and mechanistic insights. Basic Res Cardiol. 2025 Feb;120(1):35-55. doi: 10.1007/s00395-024-01034-4. Epub 2024 Feb 14. PMID 38353711
- [Result] Adams V, Reich B, Uhlemann M, Niebauer J. Molecular effects of exercise training in patients with cardiovascular disease: focus on skeletal muscle, endothelium, and myocardium. Am J Physiol Heart Circ Physiol. 2017 Jul 1;313(1):H72-H88. doi: 10.1152/ajpheart.00470.2016. Epub 2017 May 5. PMID 28476924
- [Result] Ansund J, Mijwel S, Bolam KA, Altena R, Wengstrom Y, Rullman E, Rundqvist H. High intensity exercise during breast cancer chemotherapy - effects on long-term myocardial damage and physical capacity - data from the OptiTrain RCT. Cardiooncology. 2021 Feb 15;7(1):7. doi: 10.1186/s40959-021-00091-1. PMID 33588948
- [Result] Antunes P, Joaquim A, Sampaio F, Nunes C, Ascensao A, Vilela E, Teixeira M, Capela A, Amarelo A, Marques C, Viamonte S, Alves A, Esteves D. Effects of exercise training on cardiac toxicity markers in women with breast cancer undergoing chemotherapy with anthracyclines: a randomized controlled trial. Eur J Prev Cardiol. 2023 Jul 12;30(9):844-855. doi: 10.1093/eurjpc/zwad063. PMID 36857149
- [Result] Berling-Ernst A, Yahiaoui-Doktor M, Kiechle M, Engel C, Lammert J, Grill S, Dukatz R, Rhiem K, Baumann FT, Bischoff SC, Erickson N, Schmidt T, Niederberger U, Siniatchkin M, Halle M. Predictors of cardiopulmonary fitness in cancer-affected and -unaffected women with a pathogenic germline variant in the genes BRCA1/2 (LIBRE-1). Sci Rep. 2022 Feb 21;12(1):2907. doi: 10.1038/s41598-022-06913-1. PMID 35190584
- [Result] Cardinale D, Colombo A, Bacchiani G, Tedeschi I, Meroni CA, Veglia F, Civelli M, Lamantia G, Colombo N, Curigliano G, Fiorentini C, Cipolla CM. Early detection of anthracycline cardiotoxicity and improvement with heart failure therapy. Circulation. 2015 Jun 2;131(22):1981-8. doi: 10.1161/CIRCULATIONAHA.114.013777. Epub 2015 May 6. PMID 25948538
- [Result] Fardman A, Banschick GD, Rabia R, Percik R, Fourey D, Segev S, Klempfner R, Grossman E, Maor E. Cardiorespiratory fitness and survival following cancer diagnosis. Eur J Prev Cardiol. 2021 Sep 20;28(11):1242-1249. doi: 10.1177/2047487320930873. Epub 2020 Jul 19. PMID 34551084
- [Result] Foulkes SJ, Howden EJ, Haykowsky MJ, Antill Y, Salim A, Nightingale SS, Loi S, Claus P, Janssens K, Mitchell AM, Wright L, Costello BT, Lindqvist A, Burnham L, Wallace I, Daly RM, Fraser SF, La Gerche A. Exercise for the Prevention of Anthracycline-Induced Functional Disability and Cardiac Dysfunction: The BREXIT Study. Circulation. 2023 Feb 14;147(7):532-545. doi: 10.1161/CIRCULATIONAHA.122.062814. Epub 2022 Nov 7. PMID 36342348
- [Result] Schmid P, Cortes J, Dent R, Pusztai L, McArthur H, Kummel S, Bergh J, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Untch M, Fasching PA, Cardoso F, Andersen J, Patt D, Danso M, Ferreira M, Mouret-Reynier MA, Im SA, Ahn JH, Gion M, Baron-Hay S, Boileau JF, Ding Y, Tryfonidis K, Aktan G, Karantza V, O'Shaughnessy J; KEYNOTE-522 Investigators. Event-free Survival with Pembrolizumab in Early Triple-Negative Breast Cancer. N Engl J Med. 2022 Feb 10;386(6):556-567. doi: 10.1056/NEJMoa2112651. PMID 35139274
- [Result] van der Schoot GGF, Ormel HL, Westerink NL, May AM, Elias SG, Hummel YM, Lefrandt JD, van der Meer P, van Melle JP, Poppema BJ, Stel JMA, van der Velden AWG, Vrieling AH, Wempe JB, Ten Wolde MG, Nijland M, de Vries EGE, Gietema JA, Walenkamp AME. Optimal Timing of a Physical Exercise Intervention to Improve Cardiorespiratory Fitness: During or After Chemotherapy. JACC CardioOncol. 2022 Oct 18;4(4):491-503. doi: 10.1016/j.jaccao.2022.07.006. eCollection 2022 Nov. PMID 36444224